CLINICAL TRIAL: NCT04500262
Title: Comparison Trial of Open-tip Pulsed Needle Biopsy and Conventional Core Biopsy in Axillary Lymph Nodes
Acronym: COMPULSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeoDynamics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NEODOC- 2021668610-221
Record Dates: First submitted 2020-07-22; First posted 2020-08-05 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Axillary Lymph Nodes; Biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Large-Core Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open-tip pulsed needle biopsy (Active Comparator): Biopsy procedure using the NeoNavia biopsy system. The needle used in this study is of the same outside diameter as a standard biopsy needle used in the breast or axilla (14-gauge) but does not have a notched trochar like a conventional spring-loaded device. It does not have a redundant portion of needle beyond the sampling zone and takes full circumference cylindrical cores.
  A pneumatic system powered by a floor-standing base unit connected via a handheld driver to the biopsy device provides impulses to the needle, allowing the operator to advance the needle through tissue with little manual force (NeoNavia biopsy system, NeoDynamics, Sweden).
  Interventions: Device: Open-tip pulsed needle biopsy (NeoNavia Biopsy System)
- Conventional core needle biopsy (CNB) (Active Comparator): Standard of care core needle biopsy used currently in clinics for biopsy procedures
  Interventions: Device: Core needle biopsy (CNB)

INTERVENTIONS:
Device: Open-tip pulsed needle biopsy (NeoNavia Biopsy System) — Ultrasound-guided biopsy using 14G open-tip pulsed biopsy needle
  Arms: Open-tip pulsed needle biopsy
Device: Core needle biopsy (CNB) — Ultrasound-guided biopsy using standard of care core needle biopsy
  Arms: Conventional core needle biopsy (CNB)

SUMMARY:
The aim of the study is to compare performance and safety of a newly developed 14-gauge open-tip pulsed biopsy needle with a conventional 14-gauge core biopsy needle for sampling of radiologically indeterminate or suspicious axillary lymph nodes in women with radiologically suspected breast cancer.

This is a Sponsor-initiated multicentre randomised trial. At the time of radiological breast cancer diagnosis women with ultrasonically abnormal lymph nodes undergo axillary sampling using the NeoNavia biopsy system or a common CNB device. This is in accordance with clinical routine and current clinical guidelines. The NeoNavia biopsy system is approved for use in the axillary lymph nodes.

DETAILED DESCRIPTION:
It is the standard of care in the United Kingdom for women with suspected or confirmed breast cancer to undergo ultrasound of the ipsilateral axilla prior to surgery in order to detect nodal metastatic disease. Women with invasive breast cancer and normal axillary ultrasound will then undergo operative sentinel lymph node biopsy. This is usually at the same time as the surgical removal of the breast cancer by wide local excision or mastectomy but may be done as a separate procedure before (e.g. where neoadjuvant chemotherapy is planned) or after (e.g. if a non-operative diagnosis of invasive breast cancer was not made prior to surgery). Women who are found to have a positive sentinel lymph node biopsy (i.e. have axillary metastatic disease) normally undergo axillary node clearance (ANC) at a subsequent operation. This policy may change in the future, as evidence from the American Z0011 study suggests that women with low volume axillary metastatic disease do as well with no further axillary surgery plus standard adjuvant treatment as those that undergo ANC.

Women who have abnormal lymph nodes on axillary ultrasound undergo tissue sampling with core needle biopsy (CNB), usually 14 Gauge (14G) under local anaesthetic or with fine needle aspiration cytology (FNAC). Women with proven axillary nodal metastases will then usually undergo axillary node clearance at the same operation as surgical removal of the primary tumour.

The number of women who need to undergo more than one operation can therefore be minimised by maximising the number of women with axillary metastatic disease in whom this diagnosis is made preoperatively.

Meta-analyses of published studies and more recent studies suggest that ultrasound has a sensitivity of ~60% and specificity of ~80% for the detection of metastatic lymph nodes. Although no randomised comparisons of 14G core needle biopsy (CNB) and FNAC have been performed, several studies have suggested that CNB is more accurate. Ultrasound-guided biopsy of nodes subsequently proven at surgery to contain metastases has a sensitivity of ~80% and a specificity of 100% and is more likely to be positive in those women with a higher nodal burden. Numerous studies suggest that increasing the volume of tissue removed may increase the diagnostic yield.

Recently a new biopsy device indicated for the use in breast and axillary lymph nodes (NeoNavia biopsy system, NeoDynamics, Sweden) has become available. It incorporates a pneumatic needle insertion mechanism that is intended to provide better control of needle progression and enable stepwise insertion without noticeable deformation or displacement of surrounding tissue as visualized under ultrasound. Furthermore a new method of tissue acquisition is employed that has pre-clinically shown a significantly higher sampling yield compared to CNB. These characteristics indicate that the device could be well suited for axillary lymph node biopsies. Initial clinical results indicate that in axillary lesions deemed "technically difficult", i.e. where prior US-guided biopsies with CNB or FNA had yielded non-diagnostic histology results, the NeoNavia device performed successfully, thereby significantly altering clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Women in screening and symptomatic clinics aged 18 years or older with breast masses scored as 1 of the following:

  * M3, M4 or M5 (mammographically uncertain, suspicious or highly suspicious of malignancy)
  * MRI5 (highly suspicious of malignancy on MRI)
  * U3, U4 or U5 (ultrasonically uncertain, suspicious or highly suspicious of malignancy)
  * have histologically proven breast cancer
* who have ipsilateral axillary lymph nodes which are described as indeterminate or suspicious for metastatic disease and indicated for biopsy, as determined by individual breast unit criteria
* are able to give informed consent for the study

Exclusion Criteria:

* Previous ipsilateral axillary surgery
* Target lymph node not suitable for needle biopsy due to its close proximity to critical structures such as major blood vessels
* Unable to give written informed consent in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of adequacy rate of tissue sampling of axillary lymph nodes under local anaesthetic with open-tip pulsed needle biopsy (OT-PNB) and conventional 14-gauge core needle core biopsy (CNB) | After histopathological analysis of tissue samples, up to 1 week after biopsy

SECONDARY OUTCOMES:
Comparison of pain scores for the two biopsy techniques immediately post-procedure and the maximum from days 1-3 post-procedure | 1-14 days
  Pain questionnaire administered to the participant immediately following the procedure and 4-14 days post procedure (relating to days 1-3 post procedure). Scale 0-10; 0 means no pain, 10 is the worst pain imaginable.
Comparison of complication rates between the two techniques | 0-14 days post-biopsy
  Collection of AE's, SAE's and device deficiencies
Comparison of the willingness of patients to undergo the procedure again if necessary | 4-14 days post-biopsy
  Questionnaire administered to the participant on clinic visit for biopsy result
Comparison of number of tissue samples taken with the two techniques and the number of device insertions per subject | 1 day
  Biopsy procedure data collected in real time
Comparison of the time taken for the two techniques (first biopsy device entry to last withdrawal) | 1 day
  Biopsy procedure data collected in real time
Comparison of the total weight of tissue obtained with the two techniques and the average weight per device insertion | 1 day
  Samples are weighed in clinic or pathology following the procedure
Users views upon whether the pulse technology of the NeoNavia® device facilitates accurate needle passage through the tissues to an optimum sampling position | 1 day
  Yes/No, questionnaire given to radiologist
Users views upon whether the pulse technology of the NeoNavia® device facilitates stabilisation of the target and control of the needle position | 1 day
  Yes/No, questionnaire given to radiologist
Comparison of sensitivity of preoperative axillary assessment of ultrasonically indeterminate or abnormal axillary lymph (calculated from the proportion of women with axillary metastatic disease at surgery). | post-surgery
  14-200 days
Comparison of intended outcome of biopsy procedure, i.e. number of samples to be taken from respective lymph node, and actual outcome | 1 day
  Biopsy procedure data

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Vinnicombe, Dr, Principal Investigator — Gloucestershire Hospitals NHS Foundation Trust
Locations (16):
- United Kingdom (16):
  - Basildon University Hospital, Basildon
  - Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Thirlestaine Breast Centre, Gloucestershire Hospitals NHS Foundation, Cheltenham
  - Darlington Memorial Hospital, Darlington
  - University Hospital of North Durham, Durham
  - Western General Hospital, Lothian NHS Trust, Edinburgh
  - Northwick Park Hospital, Harrow
  - High Wycombe Hospital, High Wycombe
  - Hull University Teaching Hospitals NHS Trust, Hull
  - St James's University Hospital, Leeds Teaching Hospitals NHS Trust, Leeds
  - King Edward VII's Hospital, BARTS Health NHS Trust, London
  - Wythenshawe Hospital, Manchester University NHS Foundation Trust, Manchester
  - North Manchester General Hospital, Manchester
  - Southend University Hospital, Southend
  - The Royal Marsden, The Royal Marsden NHS Foundation Trust, Sutton
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Background] Houssami N, Turner RM. Staging the axilla in women with breast cancer: the utility of preoperative ultrasound-guided needle biopsy. Cancer Biol Med. 2014 Jun;11(2):69-77. doi: 10.7497/j.issn.2095-3941.2014.02.001. PMID 25009748
- [Background] Topps AR, Barr SP, Pikoulas P, Pritchard SA, Maxwell AJ. Pre-operative Axillary Ultrasound-Guided Needle Sampling in Breast Cancer: Comparing the Sensitivity of Fine Needle Aspiration Cytology and Core Needle Biopsy. Ann Surg Oncol. 2018 Jan;25(1):148-153. doi: 10.1245/s10434-017-6090-1. Epub 2017 Oct 23. PMID 29063297
- [Background] Britton PD, Provenzano E, Barter S, Gaskarth M, Goud A, Moyle P, Sinnatamby R, Wallis M, Benson JR, Forouhi P, Wishart GC. Ultrasound guided percutaneous axillary lymph node core biopsy: how often is the sentinel lymph node being biopsied? Breast. 2009 Feb;18(1):13-6. doi: 10.1016/j.breast.2008.09.003. Epub 2008 Nov 7. PMID 18993074
- [Background] Macaskill EJ, Purdie CA, Jordan LB, Mclean D, Whelehan P, Brown DC, Evans A. Axillary lymph node core biopsy for breast cancer metastases -- how many needle passes are enough? Clin Radiol. 2012 May;67(5):417-9. doi: 10.1016/j.crad.2011.10.006. Epub 2011 Nov 26. PMID 22119100
- [Background] Maxwell AJ, Bundred NJ, Harvey J, Hunt R, Morris J, Lim YY. A randomised pilot study comparing 13 G vacuum-assisted biopsy and conventional 14 G core needle biopsy of axillary lymph nodes in women with breast cancer. Clin Radiol. 2016 Jun;71(6):551-7. doi: 10.1016/j.crad.2016.02.024. Epub 2016 Mar 31. PMID 27040801
- [Background] Giuliano AE, Hunt KK, Ballman KV, Beitsch PD, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, McCall LM, Morrow M. Axillary dissection vs no axillary dissection in women with invasive breast cancer and sentinel node metastasis: a randomized clinical trial. JAMA. 2011 Feb 9;305(6):569-75. doi: 10.1001/jama.2011.90. PMID 21304082
- [Background] POSNOC - A Trial Looking at Axillary Treatment in Early Breast Cancer (POSNOC). ClinicaltrialsGov n.d. https://clinicaltrials.gov/ct2/show/NCT02401685 (accessed February 18, 2019)
- [Background] Alvarez S, Anorbe E, Alcorta P, Lopez F, Alonso I, Cortes J. Role of sonography in the diagnosis of axillary lymph node metastases in breast cancer: a systematic review. AJR Am J Roentgenol. 2006 May;186(5):1342-8. doi: 10.2214/AJR.05.0936. PMID 16632729
- [Background] Houssami N, Ciatto S, Turner RM, Cody HS 3rd, Macaskill P. Preoperative ultrasound-guided needle biopsy of axillary nodes in invasive breast cancer: meta-analysis of its accuracy and utility in staging the axilla. Ann Surg. 2011 Aug;254(2):243-51. doi: 10.1097/SLA.0b013e31821f1564. PMID 21597359
- [Background] Joh JE, Han G, Kiluk JV, Laronga C, Khakpour N, Lee MC. Indications for axillary ultrasound use in breast cancer patients. Clin Breast Cancer. 2012 Dec;12(6):433-7. doi: 10.1016/j.clbc.2012.09.009. Epub 2012 Oct 11. PMID 23062709
- [Background] Leenders MW, Broeders M, Croese C, Richir MC, Go HL, Langenhorst BL, Meijer S, Schreurs WH. Ultrasound and fine needle aspiration cytology of axillary lymph nodes in breast cancer. To do or not to do? Breast. 2012 Aug;21(4):578-83. doi: 10.1016/j.breast.2012.05.008. Epub 2012 Jun 19. PMID 22717665
- [Background] Rattay T, Muttalib M, Khalifa E, Duncan A, Parker SJ. Clinical utility of routine pre-operative axillary ultrasound and fine needle aspiration cytology in patient selection for sentinel lymph node biopsy. Breast. 2012 Apr;21(2):210-4. doi: 10.1016/j.breast.2011.09.014. Epub 2011 Oct 5. PMID 21981897
- [Background] Garcia-Ortega MJ, Benito MA, Vahamonde EF, Torres PR, Velasco AB, Paredes MM. Pretreatment axillary ultrasonography and core biopsy in patients with suspected breast cancer: diagnostic accuracy and impact on management. Eur J Radiol. 2011 Jul;79(1):64-72. doi: 10.1016/j.ejrad.2009.12.011. Epub 2010 Jan 4. PMID 20047809
- [Background] Rao R, Lilley L, Andrews V, Radford L, Ulissey M. Axillary staging by percutaneous biopsy: sensitivity of fine-needle aspiration versus core needle biopsy. Ann Surg Oncol. 2009 May;16(5):1170-5. doi: 10.1245/s10434-009-0421-9. Epub 2009 Mar 5. PMID 19263171
- [Background] Rautiainen S, Masarwah A, Sudah M, Sutela A, Pelkonen O, Joukainen S, Sironen R, Karja V, Vanninen R. Axillary lymph node biopsy in newly diagnosed invasive breast cancer: comparative accuracy of fine-needle aspiration biopsy versus core-needle biopsy. Radiology. 2013 Oct;269(1):54-60. doi: 10.1148/radiol.13122637. Epub 2013 Jun 14. PMID 23771915
- [Background] Ganott MA, Zuley ML, Abrams GS, Lu AH, Kelly AE, Sumkin JH, Chivukula M, Carter G, Austin RM, Bandos AI. Ultrasound Guided Core Biopsy versus Fine Needle Aspiration for Evaluation of Axillary Lymphadenopathy in Patients with Breast Cancer. ISRN Oncol. 2014 Feb 4;2014:703160. doi: 10.1155/2014/703160. eCollection 2014. PMID 24649373
- [Background] van Wely BJ, de Wilt JH, Francissen C, Teerenstra S, Strobbe LJ. Meta-analysis of ultrasound-guided biopsy of suspicious axillary lymph nodes in the selection of patients with extensive axillary tumour burden in breast cancer. Br J Surg. 2015 Feb;102(3):159-68. doi: 10.1002/bjs.9663. Epub 2014 Oct 29. PMID 25354962
- [Background] Lee J, Bishop B, Allen S. NeoNavia biopsy system: Our experience of a new device for more precise ultrasound-guided percutaneous core biopsy of axillary lymph nodes. Breast Cancer Res 2017;19(suppl 1):18.
- [Background] Abe H, Schmidt RA, Sennett CA, Shimauchi A, Newstead GM. US-guided core needle biopsy of axillary lymph nodes in patients with breast cancer: why and how to do it. Radiographics. 2007 Oct;27 Suppl 1:S91-9. doi: 10.1148/rg.27si075502. PMID 18180238
- [Background] Abe H, Schmidt RA, Kulkarni K, Sennett CA, Mueller JS, Newstead GM. Axillary lymph nodes suspicious for breast cancer metastasis: sampling with US-guided 14-gauge core-needle biopsy--clinical experience in 100 patients. Radiology. 2009 Jan;250(1):41-9. doi: 10.1148/radiol.2493071483. Epub 2008 Oct 27. PMID 18955508
- See also: Schässburger et al. High velocity pulse biopsy device enables controllable and precise needle insertion and high yield tissue acquisition. Phys Med. 2018 Feb;46:25-31. doi: 10.1016/j.ejmp.2017.12.014. Epub 2018 Jan 30. — https://pubmed.ncbi.nlm.nih.gov/29519406/